CLINICAL TRIAL: NCT02751112
Title: Evaluation of a Kit for the Prediction of the Risk of Graft Versus Host Disease
Acronym: Predictor007
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment and preliminary observations leading to early termination
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IMIS2014-03
Record Dates: First submitted 2016-04-13; First posted 2016-04-26 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-08

CONDITIONS: Hemopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Couple donor / recipient (Experimental): Each couple will be treated the same way :
  An additional blood sample of the donor will be taken prior GCSF mobilization. This blood sample will then be analyzed via Predictor's kit, by the immunology laboratory of the hospital where the graft will be done.
  Whatever the result given by the Predictor' kit, the graft will be done for the recipient patient. No change will be done on the usual graft process.
  Interventions: Biological: Predictor' kit

INTERVENTIONS:
Biological: Predictor' kit — Realization of the Predictor' kit on the blood of donor of HSC, in the frame of a graft, to predict a aGvH reaction on recipient patient.

SUMMARY:
This study is a proof of concept that will assess the Predictor's kit performances. The test will be performed by several technicians, in immunological laboratories of several sites in France.

In this study, "couples" of donor / recipient in the frame of a graft of CSH will be included.

DETAILED DESCRIPTION:
The Hematopoietic Stem Cell (HSC) graft is the only curative treatment for lots of hematologic diseases, malignant or not, particularly leukemias.

The acute Graft versus Host (aGvH) reaction is the most frequent complication, and could concern until 50% of recipients. It is mainly linked to immune characteristics of the donor which will act versus the graft recipient.

There is a huge need of a technology that could predict the risk of aGvH, especially in order to select a donor in case of several possibilities, in order to reduce morbidity and mortality of graft.

The Predictor' kit allows to predict acute and severe forms of Graft versus Host disease before the graft of peripheral hematological stem cells, by the assesment of iNKT cells expansion.

ELIGIBILITY:
Main inclusion Criteria for Donors :

* Being a relative of the recipient patient, OR being registered on the National Registry of the volunteers for bone marrow donation
* Being candidate for a donation of Hematologic Stem Cells with a HLA compatibility 10/10

Main inclusion Criteria for Recipient :

* Being candidate for a donation of Hematologic Stem Cells with the following criteria:
* HLA compatibility 10/10 with the donor
* Suffering from malignant or non-malignant hemopathy in first remission
* Myeloablative or reducted intensity conditioning
* Classic scheme of immunosuppression decreasing

Main exclusion Criteria:

* Participation to a therapeutical protocol in the 30 last days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-11; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Assessment of the diagnosis test performance | 6 months
  The performance of the test will be assessed via the observation of the number of aGvH 6 months after the graft, reported to the the expansion of iNKT cells.
  Assessment of sensitivity and specificity of the diagnosis test

SECONDARY OUTCOMES:
Assessment of the reproductibility of the test | 6 months
  The reproductibility of the test will be assessed by comparing the results obtained by 2 distinct operators : the immunology lab technician, and the referent operator at Imagine Institute research lab.
  The 2 operators will perform the test in parallel on the blood of the same donor, in similar conditions, and both by using a Predictor's kit.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre Hospitalier de Caen, Caen
  - Hôpital de Huriez / CHRU de Lille, Lille
  - Hôpital Necker Enfants Malades, Paris
  - Hôpital Haut-Lévèque, Pessac